CLINICAL TRIAL: NCT04190420
Title: The Transition From Hypertension to Hypertensive Heart Disease and Heart Failure, the PREFERS Hypertension Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Mattias Ekström, Dr, Karolinska Institutet
Other Study IDs: 2019-00898
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Hypertension; Heart Failure; Hypertensive Heart Disease; Diastolic Dysfunction
Keywords: Hypertension; Hypertensive heart disease; Heart failure; Biomarkers; Diastolic dysfunction
MeSH Terms: conditions — Hypertension; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For future analysis of biomarkers and DNA extraction, aliquots of whole blood, plasma and serum will be stored in freezers (-80 degrees C) in the Stockholm Medical Biobank (Bbk2132) until analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: 250 patients with primary hypertension
- Healthy Controls: 60 healthy control subjects, matched in age and gender

SUMMARY:
AIMS Despite evidence-based therapeutic approaches, target blood pressure is obtained by less than half of patients with hypertension. Hypertension is associated with a significant risk for heart failure (HF), in particular HF with preserved left ventricular (LV) ejection fraction (HFpEF). Although treatment is suggested to be given early after hypertension diagnosis, there is still no evidence-based medical treatment for HFpEF. We aim to study the underlying mechanisms behind the transition from uncomplicated hypertension to hypertensive heart disease (HHD) and HFpEF. To this end, we will combine cardiac imaging techniques and measurements of circulating fibrosis markers to longitudinally monitor fibrosis development in patients with hypertension.

METHODS In a prospective cohort study, 250 patients with primary hypertension and 60 healthy controls, will be characterized at inclusion, and after 1 and 6 years. Doppler-echocardiography, cardiac magnetic resonance imaging (CMR) and ECG will be used for measures of cardiac structure and function over time. Blood biomarkers reflecting myocardial fibrosis, inflammation and endothelial dysfunction will be analysed. As a proxy for HFpEF development, the primary endpoint is to measure echocardiographic changes in LV function and structure (E/e´ and LAVI) and to relate these measures of LV filling to blood pressure, biomarkers, ECG and CMR.

CONCLUSION We aim to study the timeline and transition from uncomplicated hypertension to HHD and HFpEF. In order to identify subjects prone to develop HHD and HFpEF, we want to find biomarkers and cardiac imaging variables to explain disease progression. Ultimately, we aim at finding new pathways to prevent HFpEF.

DETAILED DESCRIPTION:
INTRODUCTION Hypertension is common with a prevalence of approximately one third of the adult Swedish population and similar figures reported world wide. It is associated to cardiac structural- and functional changes as well as vascular dysfunction which all can be delayed or reversed by appropriate antihypertensive treatment. Although blood pressure (BP) control is improving, target BP is still reached by less than half of the treated patients. Hypertension is the single risk factor with the greatest attributable risk for incident heart failure (HF) and is considerably more common in HF with preserved left ventricular (LV) ejection fraction (HFpEF) than in HF with reduced EF (HFrEF). In patients with established HFpEF hypertension is very common, ranging between 50-70%. However, the exact mechanisms for the transition from hypertension to hypertensive heart disease and HFpEF are less well understood. In contrast, pathophysiology and progression of HFrEF is better elucidated and may successfully be reversed by 7-8 evidence-based treatments.

The evolution of myocardial fibrosis may be one early important mechanism in the transition from hypertension to HHD, and subsequent heart failure. This can be studied through the recent development of cardiac imaging with advanced Doppler-echocardiography, cardiac magnetic resonance (CMR) imaging, and assessment of circulating biomarkers reflecting myocardial fibrosis turnover, inflammation and endothelial dysfunction. Indeed, echocardiographic left chamber longitudinal strain and extracellular volume measured by CMR have recently been demonstrated to be useful to discriminate between healthy controls, patients with hypertension and patients with HFpEF. Also circulating plasma biomarkers reflecting altered myocardial tissue turnover can differentiate patients with left ventricular hypertrophy (LVH) from patients with LVH and HFpEF. In addition, biomarkers may identify phenotypes of high collagen cross-linking which has been suggested to have impact on the response to medical treatment in HFpEF.

An increased understanding of these mechanisms allows the development of specific treatments, guided by cardiac imaging and/or biomarker assessments, to delay or prevent the transition from hypertension to HF. This may have considerable clinical implications in reducing cardiovascular complications to hypertension. Thus, the aim of the present study is to characterize and study the timeline and the transition from uncomplicated hypertension to HHD and HFpEF in subjects with primary hypertension using advanced cardiac imaging techniques and bioinformatics, Table 1. Furthermore, we aim to compare changes of HFpEF variables and biomarkers in this study to patients with new onset symptomatic HFpEF in the Stockholm PREFERS Heart failure study, see below.

Table 1.

HYPOTHESES:

1. Hypertension with normal left atrial/ventricular function deteriorates over time, starting with increasing filling pressure, left atrial enlargement followed by reduced global longitudinal strain with LVEF>50% and heart failure symptoms (HFpEF)
2. Circulating biomarkers reflecting myocardial fibrosis, inflammation and endothelial dysfunction reflects the transition from hypertension to hypertensive heart disease and HFpEF

As a proxy for HFpEF development our OVERALL AIM is to investigate:

if change in diastolic cardiac function E/e' or left atrial volume index (LAVI) after one year is associated to blood pressure at baseline.

SPECIFIC AIMS:

1. to study if change in diastolic cardiac function measured with E/e' or LAVI after one year is associated to change in blood pressure from baseline to one year.
2. to assess if blood pressure control at baseline (according to guidelines and age adjusted) is associated to diastolic cardiac function measured with E/e' or LAVI after one year.
3. to investigate if blood pressure control after one year (according to guidelines and age adjusted) is associated to diastolic cardiac function measured with E/e' or LAVI after one year.
4. to study the temporal evolution (baseline, one year, six years) of the diastolic function measured with E/e' or LAVI.
5. to investigate gender aspects on the temporal evolution (baseline, one year, six years) of the diastolic function measured with E/e' or LAVI.
6. to study the temporal evolution (baseline, one year, six years) of the diastolic function measured with echocardiography and CMR.
7. to assess if temporal changes (baseline, one year, six years) in circulating levels of biomarkers reflecting myocardial fibrosis, inflammation and endothelial dysfunction are associated with changes in blood pressure.
8. to assess if temporal changes (baseline, one year, six years) in circulating levels of biomarkers reflecting myocardial fibrosis, inflammation and endothelial dysfunction are associated with changes in diastolic function.

METHODS

STUDY DESIGN The study PREFERS Hypertension, is the last part of the PREFERS (Preserved and Reduced Ejection Fraction Epidemiological Regional Study in Stockholm, Clin trial NCT03671122), a clinical trial first aiming at describing underlying pathophysiological mechanisms in new onset HF, either HFpEF or HFrEF with approximately 600 patients. PREFERS Hypertension study is a single-centre, prospective clinical cohort study performed in collaboration between the Department of Cardiology at Danderyd Hospital and the Primary Health Care Services in Stockholm, Sweden. The study will recruit patients with a diagnosis of primary hypertension with an ongoing antihypertensive drug treatment as well as healthy control subjects, for comparison as previously described. For inclusion and exclusion criteria, see below. All subjects will be assessed at the Cardiovascular Research Laboratory, which is part of the Clinical Research Centre at Danderyd University Hospital.

Primary hypertension is defined as a diagnosis documented in primary care at some time point within the last 24 months and ongoing antihypertensive drug treatment (maximum up to 2-3 drugs). The currently recommended definition of hypertension as a systolic office BP >140 mmHg and/or diastolic BP >90 mmHg(19) is widely adapted in primary health care. Exclusion of secondary hypertension is at the discretion of the primary health care physician or may be excluded at the inclusion visit. Controlled hypertension is defined as <140/90 mm Hg.

RECRUITMENT OF STUDY PARTICIPANTS AND TIMELINE Hypertension in Sweden is usually managed at primary health care centers. Through a collaboration between hospital and primary care, the patients will be recruited from health care centers in various socioeconomic areas in Stockholm (approximately 10 care centers, total catchment area of 100 000 inhabitants). To include 250 patients and with an expected response rate of 25-30%, each health care center will identify and randomly select and invite 100 patients, gender 1:1 using the software MedRave4 (Medrave Software AB, Stockholm, Sweden). Patients will be characterized at baseline, after 1 and 6 years per standardized protocol, and they will have their medication optimized at baseline and follow-ups, according to ESC/ESH 2018 guidelines. Parallel with patient recruitment, healthy control subjects, matched in age and gender will be recruited by advertisement in local newspapers. Inclusion will be performed following a telephone interview, confirming they are apparently healthy and have no daily medication. Control subjects will follow the same study protocol as the patients but planned to be examined at inclusion only. The study protocol has been approved by the regional Ethics committee and the Stockholm Health Care services, and all study participants will give their written informed consent.

MEASUREMENTS All study data will be collected into electronic case report forms (eCRF) using the Research Electronic Data Capture (REDCap).

BLOOD PRESSURE MEASUREMENTS AND PULSE WAVE VELOCITY Seated BP measurements will be made in accordance to current ESC/ESH 2018 guidelines. Three consecutive BP measurements are recorded, 1-2 min apart, using an oscillometry device (Omron M3 Comfort, OMROM Healthcare Co., Ltd. Kyoto, Japan). BP will also be measured 1 min and 3 min after standing from a seated position, to assess orthostatic hypotension. To screen for lower extremity artery disease an ankle-brachial index will be recorded, using continuous wave Doppler.

Ambulatory blood pressure monitoring (ABPM) during 24 h will be assessed by a Spacelabs ABP monitoring 90217A device (Spacelabs Healthcare, Snoqualmie, WA, US), programmed to record BP at 20 min intervals to provide an average BP value for day-time, night-time and 24h. A diary of the patients´ activities and sleep-time will be recorded. A minimum of 70% useable BP recordings are required for a valid ABPM session. The diagnostic threshold for hypertension is according to ESC/EHS 2018 guidelines. The carotid-femoral pulse wave velocity (PWV) is assessed by the SphygmoCor XCEL device (AtCor Medical, Sydney, Australia), which allows for non-invasive assessment of the central arterial pressure waveform and measures of aortic stiffness.

ELECTROCARDIOGRAM 12 lead ECG data will be stored digitally (EC store version 4.1; Cardiolex Medical AB, Stockholm, Sweden). In harmony with the PREFERS HF study, LVH will be assessed according to the Sokolov Lyon index. In addition, beside a conventional 12-lead ECG we will analyse a resting 12-lead ECG that combines advanced and conventional ECG parameters within computerized ECG-scores which have been demonstrated to increase the detection accuracy of concentric LVH and in screening for LV systolic dysfunction.

ECHOCARDIOGRAPHIC AND CMR MEASUREMENTS We will follow current recommendations for echocardiography to record two-dimensional echocardiographic and Doppler variables, and perform Doppler tissue imaging similar to those measured in the PREFERS HF study. All measurements will be presented as mean values of three cardiac cycles. A Vivid E9 (GE, Waukesha, Wisconsin, USA) Ultrasound System will be used. To reduce interobserver variability only two sonographers will perform the investigations, which will be stored on a digital server, and will be analyzed offline.

For CMR, a Siemens Aera system (Siemens Healthcare, Erlangen, Germany) will be used to deliver standard measurements of chamber dimensions and function, and signs of tissue scars of ischemic and non-ischemic origin. Myocardial extracellular matrix and signs of fibrosis will be examined by T1 mapping. Fully automated quantitative perfusion mapping during rest and adenosine stress will give a quantitative measurement for perfusion in mL/min/g, which will be used to search for perfusion defects; both focal defects due to obstructive coronary artery disease and defects in the global myocardial perfusion reserve due to coronary microvascular disease.

MEASUREMENTS QUESTIONNAIRES Quality of life measurements are to be assessed with validated instruments; the EuroQol-5 dimensions (EQ-5D), the Kansas City cardiomyopathy questionnaire (KCCQ-12) and the Minnesota living with heart failure questionnaire (MLHFQ). To screen for excessive daytime sleepiness, we will use the Epworth Sleepiness Scale (ESS) version 1.0.

SCREENING FOR OBSTRUCTIVE SLEEP APNEA Screening for sleep disorders and obstructive sleep apnea (OSA) is performed at inclusion by the Somnocheck micro CARDIO (Weinman, Hamburg, Germany), self-applied by the study participants at home before bedtime. The ambulatory overnight cardio-respiratory polygraphy recording will measure apnea/hypopnea-, desaturation- and arousal indices.

PERIPHERAL VENOUS BLOOD- AND URINE SAMPLING Peripheral blood and urine will be collected after overnight fasting with no ingestion of caffeine or nicotine within at least 12h. Clinical routine analyses of plasma and urine will be performed directly, but for future analysis of biomarkers and DNA extraction, aliquots of whole blood, plasma and serum will be stored at -80 degrees C in the Stockholm Medical Biobank until further analysis. This ensures a standardized handling of biomaterial with high security and traceability also for long-term storage. In the PREFERS Hypertension study we plan to analyze the same panel of biomarkers as for the PREFERS HF study(17), which will enable a comparison between the two cohorts. Here, we focus on biomarkers indicative of various pathophysiological mechanisms relevant to HFpEF, including those reflecting myocardial fibrosis, inflammation and endothelial dysfunction. Fibrosis i.e: Collagen split products PICP, CITP-I, sST2, Galectin-3, MMPs and IGFBP2; Inflammation i.e: HsCRP, IL-6, E-selectin, TNF-alfa, YLK-40, GDF15; Endothelial dysfunction i.e: ICAM-1, VCAM-1, Allantoin, SDMA, ADMA, Calprotectin, Arginin, von Willebrand factor, EMPs.

OUTCOME MEASURES Mortality data outside hospital and incident admission to hospital due to heart failure will be obtained by merging the Swedish cause of death register and the Swedish national inpatient register. The unique personal identification number of all Swedish citizens will ascertain complete follow-up.

PRIMARY ENDPOINT AND STATISTICAL POWER As a proxy for HFpEF development our overall aim is to investigate if change in diastolic cardiac function E/e' or left atrial volume index (LAVI) after one year is associated to blood pressure at baseline. Therefore, the primary endpoint in this study is, either mean change of E/e' of 2 or more, or mean change of LAVI of 4 mL/m2 or more after one year. These assumptions are based on a cross-sectional analysis of a big cohort from Olmsted County, Minnesota, where clear-cut differences were shown for these echocardiographic variables in patients with hypertension, HFpEF and healthy controls. To reach 80% power at a 2-sided level of significance of 0.05 the present study is planned to recruit 250 patients and 60 healthy controls, including 20% drop outs.

ELIGIBILITY:
Inclusion Criteria:

* Primary hypertension
* Age ≥ 18 years
* Preserved cognitive function and expected longevity 1 year
* Written informed consent

Exclusion Criteria:

* Heart failure and/or reduced LVEF
* Valvular heart disease of hemodynamic importance
* Resistant hypertension
* Pregnancy
* Renal failure, GFR <30 mL/min/1,73 m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with primary hypertension will be recruited from health care centers in various socioeconomic areas in Stockholm. To include 250 patients and with an expected response rate of 25-30%, each health care center will identify and randomly select and invite 100 patients, gender 1:1. Patients will be characterized at baseline, after 1 and 6 years per standardized protocol and they will have their medication optimized at baseline and follow-ups, according to guidelines. Parallel with patient recruitment, healthy control subjects, matched in age and gender will be recruited by advertisement in local newspapers. Inclusion will be performed following a telephone interview, confirming they are apparently healthy and have no daily medication. Control subjects will follow the same study protocol as the patients but planned to be examined at inclusion only.
Sampling Method: Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Overall Aim | one year
  if change in diastolic cardiac function E/e' or left atrial volume index (LAVI) after one year is associated to blood pressure at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Ekström, Dr, Principal Investigator — Karolinska Institutet
Locations (1):
- Mattias Ekström, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
The regional ethics committee has not approved any sharing of individual participant data. If this question comes up later we have to write a new application för ethical approval but still, all data has to be coded and pseudonymized.

REFERENCES:
- [Background] Lindholm L, Agenäs I, Carlbeg B, Dahlgren H, de Faire U, Hedblad B, et al. Moderately elevated blood pressure. A systematic literature review. The Swedish Council on Technology Assessment in Health Care SBU-rapport 2004;170/1-2.
- [Background] NCD Risk Factor Collaboration (NCD-RisC). Worldwide trends in blood pressure from 1975 to 2015: a pooled analysis of 1479 population-based measurement studies with 19.1 million participants. Lancet. 2017 Jan 7;389(10064):37-55. doi: 10.1016/S0140-6736(16)31919-5. Epub 2016 Nov 16. PMID 27863813
- [Background] Jekell A, Nilsson PM, Kahan T. Treatment of Hypertensive Left Ventricular Hypertrophy. Curr Pharm Des. 2018;24(37):4391-4396. doi: 10.2174/1381612825666181203092918. PMID 30501597
- [Background] Holmquist C, Hasselstrom J, Bengtsson Bostrom K, Manhem K, Wettermark B, Hjerpe P, Kahan T. Improved treatment and control of hypertension in Swedish primary care: results from the Swedish primary care cardiovascular database. J Hypertens. 2017 Oct;35(10):2102-2108. doi: 10.1097/HJH.0000000000001429. PMID 28582282
- [Background] Levy D, Larson MG, Vasan RS, Kannel WB, Ho KK. The progression from hypertension to congestive heart failure. JAMA. 1996 May 22-29;275(20):1557-62. PMID 8622246
- [Background] Lee DS, Gona P, Vasan RS, Larson MG, Benjamin EJ, Wang TJ, Tu JV, Levy D. Relation of disease pathogenesis and risk factors to heart failure with preserved or reduced ejection fraction: insights from the framingham heart study of the national heart, lung, and blood institute. Circulation. 2009 Jun 23;119(24):3070-7. doi: 10.1161/CIRCULATIONAHA.108.815944. Epub 2009 Jun 8. PMID 19506115
- [Background] Donal E, Lund LH, Oger E, Hage C, Persson H, Reynaud A, Ennezat PV, Bauer F, Sportouch-Dukhan C, Drouet E, Daubert JC, Linde C; KaRen Investigators. Baseline characteristics of patients with heart failure and preserved ejection fraction included in the Karolinska Rennes (KaRen) study. Arch Cardiovasc Dis. 2014 Feb;107(2):112-21. doi: 10.1016/j.acvd.2013.11.002. Epub 2013 Dec 30. PMID 24388161
- [Background] Lam CS, Donal E, Kraigher-Krainer E, Vasan RS. Epidemiology and clinical course of heart failure with preserved ejection fraction. Eur J Heart Fail. 2011 Jan;13(1):18-28. doi: 10.1093/eurjhf/hfq121. Epub 2010 Aug 3. PMID 20685685
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Nagueh SF, Smiseth OA, Appleton CP, Byrd BF 3rd, Dokainish H, Edvardsen T, Flachskampf FA, Gillebert TC, Klein AL, Lancellotti P, Marino P, Oh JK, Alexandru Popescu B, Waggoner AD; Houston, Texas; Oslo, Norway; Phoenix, Arizona; Nashville, Tennessee; Hamilton, Ontario, Canada; Uppsala, Sweden; Ghent and Liege, Belgium; Cleveland, Ohio; Novara, Italy; Rochester, Minnesota; Bucharest, Romania; and St. Louis, Missouri. Recommendations for the Evaluation of Left Ventricular Diastolic Function by Echocardiography: An Update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. Eur Heart J Cardiovasc Imaging. 2016 Dec;17(12):1321-1360. doi: 10.1093/ehjci/jew082. Epub 2016 Jul 15. No abstract available. PMID 27422899
- [Background] Webb J, Fovargue L, Tondel K, Porter B, Sieniewicz B, Gould J, Rinaldi CA, Ismail T, Chiribiri A, Carr-White G. The Emerging Role of Cardiac Magnetic Resonance Imaging in the Evaluation of Patients with HFpEF. Curr Heart Fail Rep. 2018 Feb;15(1):1-9. doi: 10.1007/s11897-018-0372-1. PMID 29404975
- [Background] Gyongyosi M, Winkler J, Ramos I, Do QT, Firat H, McDonald K, Gonzalez A, Thum T, Diez J, Jaisser F, Pizard A, Zannad F. Myocardial fibrosis: biomedical research from bench to bedside. Eur J Heart Fail. 2017 Feb;19(2):177-191. doi: 10.1002/ejhf.696. PMID 28157267
- [Background] Paulus WJ, Tschope C. A novel paradigm for heart failure with preserved ejection fraction: comorbidities drive myocardial dysfunction and remodeling through coronary microvascular endothelial inflammation. J Am Coll Cardiol. 2013 Jul 23;62(4):263-71. doi: 10.1016/j.jacc.2013.02.092. Epub 2013 May 15. PMID 23684677
- [Background] Mordi IR, Singh S, Rudd A, Srinivasan J, Frenneaux M, Tzemos N, Dawson DK. Comprehensive Echocardiographic and Cardiac Magnetic Resonance Evaluation Differentiates Among Heart Failure With Preserved Ejection Fraction Patients, Hypertensive Patients, and Healthy Control Subjects. JACC Cardiovasc Imaging. 2018 Apr;11(4):577-585. doi: 10.1016/j.jcmg.2017.05.022. Epub 2017 Aug 16. PMID 28823736
- [Background] Zile MR, Desantis SM, Baicu CF, Stroud RE, Thompson SB, McClure CD, Mehurg SM, Spinale FG. Plasma biomarkers that reflect determinants of matrix composition identify the presence of left ventricular hypertrophy and diastolic heart failure. Circ Heart Fail. 2011 May;4(3):246-56. doi: 10.1161/CIRCHEARTFAILURE.110.958199. Epub 2011 Feb 24. PMID 21350055
- [Background] Ravassa S, Trippel T, Bach D, Bachran D, Gonzalez A, Lopez B, Wachter R, Hasenfuss G, Delles C, Dominiczak AF, Pieske B, Diez J, Edelmann F. Biomarker-based phenotyping of myocardial fibrosis identifies patients with heart failure with preserved ejection fraction resistant to the beneficial effects of spironolactone: results from the Aldo-DHF trial. Eur J Heart Fail. 2018 Sep;20(9):1290-1299. doi: 10.1002/ejhf.1194. Epub 2018 Apr 30. PMID 29709099
- [Background] Linde C, Eriksson MJ, Hage C, Wallen H, Persson B, Corbascio M, Lundeberg J, Maret E, Ugander M, Persson H; Stockholm County/Karolinska Institutet 4D heart failure investigators. Rationale and design of the PREFERS (Preserved and Reduced Ejection Fraction Epidemiological Regional Study) Stockholm heart failure study: an epidemiological regional study in Stockholm county of 2.1 million inhabitants. Eur J Heart Fail. 2016 Oct;18(10):1287-1297. doi: 10.1002/ejhf.599. Epub 2016 Jul 7. PMID 27384611
- [Background] Lam CS, Roger VL, Rodeheffer RJ, Bursi F, Borlaug BA, Ommen SR, Kass DA, Redfield MM. Cardiac structure and ventricular-vascular function in persons with heart failure and preserved ejection fraction from Olmsted County, Minnesota. Circulation. 2007 Apr 17;115(15):1982-90. doi: 10.1161/CIRCULATIONAHA.106.659763. Epub 2007 Apr 2. PMID 17404159
- [Background] Williams B, Mancia G, Spiering W, Agabiti Rosei E, Azizi M, Burnier M, Clement DL, Coca A, de Simone G, Dominiczak A, Kahan T, Mahfoud F, Redon J, Ruilope L, Zanchetti A, Kerins M, Kjeldsen SE, Kreutz R, Laurent S, Lip GYH, McManus R, Narkiewicz K, Ruschitzka F, Schmieder RE, Shlyakhto E, Tsioufis C, Aboyans V, Desormais I; ESC Scientific Document Group. 2018 ESC/ESH Guidelines for the management of arterial hypertension. Eur Heart J. 2018 Sep 1;39(33):3021-3104. doi: 10.1093/eurheartj/ehy339. No abstract available. PMID 30165516
- [Background] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2015 Jan;28(1):1-39.e14. doi: 10.1016/j.echo.2014.10.003. PMID 25559473